CLINICAL TRIAL: NCT06990906
Title: BENCHMARK SPERM: A Prospective, Randomized Controlled Study Evaluating the Safety and Clinical Efficacy of the BAIBYS™ System in Intracytoplasmic Sperm Injection (ICSI)
Brief Title: Evaluating the Safety and Clinical Efficacy of the BAIBYS™ System in Intracytoplasmic Sperm Injection (ICSI)
Acronym: Benchmark
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BAIBYS Fertility (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLN-009
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Male Infertility, Azoospermia
Keywords: ICSI; ART; Oocyte; Spermatozoa; Blastocyst
MeSH Terms: conditions — Infertility, Male; Azoospermia

STUDY DESIGN:
Intervention Model Description: Software-based decision support automated device for ideal sperm selection for ICSI
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- BAIBYS+ICSI treatment arm (Experimental): Oocytes of this group will be fertilized with sperm selcted by the BAIBYS System
  Interventions: Device: BAIBYS Sperm selection; Procedure: Intra cytoplasmatic sperm injection; Procedure: Conventional manual sperm selection
- ICSI control arm (Active Comparator): Oocytes of this group will be fertilized with sperm selcted by conventional manual procedre
  Interventions: Procedure: Intra cytoplasmatic sperm injection; Procedure: Conventional manual sperm selection

INTERVENTIONS:
Device: BAIBYS Sperm selection — Software based decision support device for sperm selction based on morphology and motility
  Arms: BAIBYS+ICSI treatment arm
Procedure: Intra cytoplasmatic sperm injection — Sperm injection into oocytes for ferilization
Procedure: Conventional manual sperm selection — selection beased on motility at low magnification

SUMMARY:
This study looks at an investigational automated, artificial intelligence (AI)-based sperm selection technology called the BAIBYS™ System. We want to see how it compares to current methods in terms of efficiency and effectiveness in producing high-quality Embryos, which can lead to successful pregnancies and healthy babies.

Infertility impacts about 15% of couples globally, with male issues contributing to around 50% of these cases. You will be undergoing a treatment called Intra-Cytoplasmic Sperm Injection (ICSI) as part of your planned treatment program. In this procedure, embryologists inject selected sperm into an egg, based on its movement, observed under a low-magnification microscope. However, this method does not fully detect defects in sperm shape that may indicate sperm quality. Recent studies show that using high magnification for sperm selection is important for successful fertilization, higher embryo quality, lower birth defect rates, and higher birth rates of healthy babies.

Selecting sperm manually under a microscope at high magnification takes a lot of time and depends on the skill of embryologists, which can lead to differences in judgment. Because of this, there is an interest in using AI to make sperm selection more accurate, consistent, and faster.

The BAIBYS™ System uses advanced AI technology to automatically choose sperm based on their movement, size, and shape. These features help to determine the sperm's potential to be normal and produce a good embryo. The system also organizes the selected sperm into separate areas from which the embryologist will pick the sperm for injection into the egg. This investigational device could become a valuable tool in reproductive technology. Clinical research is crucial to confirm these ideas and show their long-term effects on fertility treatments.

In this study, half of the oocytes retrieved during your IVF cycle will be injected with sperm selected from your partner's (or known donor's) semen by using the BAIBYS™ System, while the other half will be fertilized by sperm chosen according to the standard procedure at this institution. In any case, the embryologist will confirm that the sperm selected by the device are viable and acceptable. After fertilization, the best embryo, no matter which study group, will be selected for transfer to the uterus for pregnancy, and the rest of the good embryos will be frozen based on the institution's best standard clinical guidelines.

DETAILED DESCRIPTION:
The BAIBYS™ System is an automated microscopy-based tool intended to assist embryologists in selecting ideal spermatozoa based on morphological characteristics and motility for the Intra Cytoplasmic Sperm Injection (ICSI) procedure. It employs computer-vision machine learning algorithms trained with high-magnification live cell imagery. The system is indicated for adults who are undergoing the ICSI procedure.

Prospective, multi-center, two-arms (standard ICSI+BAIBYS™ vs. Standard ICSI only) randomized controlled study.

* The sperm selection methodology utilized in the BAIBYS™ System for ICSI serves as a software-based decision-support tool. The embryologist retains the final decision regarding the utilization of the sperm that has been chosen by the apparatus.
* The determination of the selected embryo for transferring to the uterine cavity and cryopreservation is based on the best conventional clinical practice. The study design directs only in cases of multiple decision options in order to maintain the balance between the sample size of the study cohorts.
* Each female participant will be equally randomized to either the BAIBYS™ arm or the Control arm. This randomization will determine the oocyte (extra) allocation, ICSI timing, and embryo transfer:

  * The extra oocyte in case of an odd number will be assigned to the arm per the randomization plan
  * The injection of spermatozoa from both arms will be administered as close as possible. Priority will be given according to the randomization plan.
  * The embryo designated for transfer into the uterus will be selected based on the randomization plan in case the two best embryos from different arms exhibit similar quality assessment grading.
* The embryologists who inject sperm into the oocytes of both arms will remain blind to the study arm from which the sperm originated. The selected sperm in each arm will be transferred to a new ICSI dish in which the allocated oocytes are placed.

ELIGIBILITY:
Inclusion Criteria:

1. Couples intended to be ICSI recruited from the clinic's IVF units. Couples may be utilizing their own gametes, or gametes from one known donor (for donated gametes, the donor will also need to consent).
2. Male subject aged ≥ 21 years at the time of screening
3. Male subjects with at least 1 abnormal parameter at the sperm analysis according to the WHO criteria (count, motility, or morphology)
4. Female subjects aged 21 to 42 years at the time of screening
5. Number of follicles ≥14 mm as measured by ultrasound evaluation at ovulation trigger is at least 11
6. The subject can provide a sperm sample by ejaculation. Sperm can be produced by electric ejaculation. Fresh or thawed sperm can be used for the procedure.
7. Total Motile sperm Count (TMC) > 1 million
8. The subject can understand and sign a written informed consent form

Exclusion Criteria:

1. Severe grade IV endometriosis (suspected or confirmed by surgery), moderate to severe adenomyosis, or a condition that is known to render implantation unlikely, such as 3 or more prior losses related to uterine issues.
2. Sperm produced by TESE (testicular sperm extraction)/TESA (testicular sperm aspiration).
3. The subjects are under active oncology treatment.
4. Participation in another study with any investigational drug or device that may conflict with the objectives, follow-up, or testing of this study.
5. Planned sex selection or any other scenario where a less-optimal embryo is planned to be transferred
6. Anonymous donor or other donor scenarios where it is uncertain whether freely given consent can be obtained

Ages: 21 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Co-primary: Usable Blastocyte formation rate and Clinical Pregnancy rate | 5-6 days post ICSI and 7 weeks post embryo transfer
  A co-primary clinical performance endpoint.
  1. Usable Blastocyst Rate Using Gardner's scoring, a superiority margin of 5% between the BAIBYS™ treatment arm and the standard ICSI arm of usable blastocyst development rate (≥3BB) at day 5 or 6 post-insemination (Embryos that do not reach the blastocyst stage by day 5 but continue to develop into morulae or blastocysts shall be followed and reassessed on day 6).
  2. Clinical Pregnancy Rate A superiority margin of 1% between the BAIBYS™ treatment arm and the standard ICSI arm of the proportion of embryo transfers resulting in a clinical pregnancy confirmed at week 7±1 by ultrasound visualization of an intrauterine gestational sac with fetal heartbeat
Irreversible SADE | 1-day post-ICSI
  The incidence of irreversible Serious Adverse Device (SADE) in the BAIBYS™ treated arm group is ≤ 5%.
  Incidence encompasses deficiencies associated with the device, including user error, device malfunction, or suboptimal performance resulting in the incapacity to effectively and safely execute the ICSI procedure

SECONDARY OUTCOMES:
Procedure Efficiency | ICSI day 0
  The median time for selection of a spermatozoon by the BAIBYS™ System is ≤ 3 minutes
Pregnancy rate | 6-8 weeks post embryo transfer
  The rate of clinical pregnancy in weeks 6-8, as indicated by the presence of a normal heartbeat, within the BAIBYS™ treatment cohort transferred embryos is ≥ 35% or is at least 5% higher than in the standard ICSI treatment cohort
Fertilization rate | 16-18 hours post-ICSI
  The rate of oocyte fertilization within the BAIBYS™ treatment cohort (defined as the proportion of oocytes exhibiting two pronuclei or undergoing cellular division at 16-18 hours post-ICSI) exceeds 65% or is at least 5% higher than in the standard ICSI treatment cohort

OTHER OUTCOMES:
Blastocyte formation rate as a function of 2PN zygote | 5-6 days post ICSI
  A comparative analysis of the proportion of usable blastocyte development on day 5/6 as a function of 2PN zygote across both study arms
Implantation rate | 1 day post embryo transfer
  A comparative analysis of the proportion of successful implantation across both study arms
Biochemistry pregnancy rate | 12 to 14 post-embryo transfer
  A comparative analysis of the proportion of pregnancy, as indicated by the presence of positive HCG on days 12 to 14 post-embryo transfer across both study arms

CONTACTS AND LOCATIONS:
Locations (3):
- New England Fertility Institute, Stamford, Connecticut, United States
- Assuta Medical Center, Tel Aviv, Israel
- Care Fertility Group, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No